CLINICAL TRIAL: NCT07399418
Title: TRIAD - Tracking Risk in Integrated Alzheimer's Diagnostics. A Biopsychosocial Model for the Early and Accurate Diagnosis of the Alzheimer's Disease Continuum.
Brief Title: TRIAD - Tracking Risk in Integrated Alzheimer's Diagnostics.
Acronym: TRIAD
Status: Recruiting | Type: Observational
Sponsor: Istituti Clinici Scientifici Maugeri SpA (Other)
Collaborators: Catholic University of the Sacred Heart (Other); Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-3.11/337
Record Dates: First submitted 2026-01-20; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Cognitive Decline
Keywords: Alzheimer's disease; Early diagnosis; Cognitive impairment; Biopsychosocial model; Caregiver; Neuropsychological rehabilitation; Mild cognitive impairment; Subjective cognitive decline; blood biomarkers
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease; Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood biomarkers of neurodegeneration, including: the peptide β-amyloid 40 (Aβ40), β-amyloid 42 (Aβ42), phosphorylated tau at position 181 (p-Tau181), and neurofilament light chain (NfL) u Blood biomarkers of neuroinflammation, including: glial fibrillary acidic protein (GFAP), soluble receptor for activation expressed on myeloid cells 2 (sTREM2), and chitinase-3-like protein 1 (YKL40).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study is based on the hypothesis that the integration of biological, psychological, and social factors, according to the biopsychosocial paradigm, allows for more accurate identification of the different stages of the Alzheimer's continuum (AD), facilitating early diagnosis and effective management. It is also hypothesized that the experience of the caregiver is a key element, capable of influencing the patient's experience and clinical course, representing a potential early indicator of risk.

Primary objectives are (PO.1) Jointly analyze biological, psychological, and social factors at different stages of the AD continuum to construct multidimensional clinical profiles and integrated risk models.

(PO.2) Examine the influence of psychological and social variables on the quality of life of patients and caregivers at different stages of the disease.

(PO.3) Investigate the relationship between caregiver psychological well-being and patient cognitive functioning, exploring potentially bidirectional relationships.

Secondary objectives are (SO.1) Compare biomarkers and neuropsychological performance at different stages of the AD clinical continuum.

(SO.2) Evaluate the diagnostic effectiveness of blood and neuroimaging biomarkers in discriminating the severity of cognitive impairment.

(SO.3) Explore stress and coping strategies adopted by caregivers, in relation to the stage of the disease and the quality of the dyadic relationship.

(So.4) Integrate quantitative and qualitative data to understand the emotional experience of the caregiver throughout the entire disease continuum.

DETAILED DESCRIPTION:
Background

Global aging is leading to an increase in the prevalence of dementia, with an estimated 50 million cases worldwide. Among these, Alzheimer's disease (AD) is the most widespread, characterized by a progressive neurodegenerative course with cognitive, behavioral, and functional symptoms. AD is now considered a pathological continuum with six progressive stages, where the first two, preclinical stages represent a crucial window for early intervention. However, diagnostic methods such as CSF and PET, although effective, are expensive and invasive. Recent research suggests that blood biomarkers of neuroinflammation could offer more accessible solutions.

Understanding the early stages of AD is complicated by their subjectivity, making the use of a purely biomedical model insufficient. The biopsychosocial paradigm integrates biological, psychological, and social aspects, offering a more comprehensive view of the disease. In this context, the role of the caregiver is also central. As AD progresses, the patient becomes dependent, with a direct impact on the quality of life and mental health of the caregiver, who often experiences stress, anxiety, and depression. Work and relationship difficulties increase the emotional and caregiving burden, making it important to consider the caregiver's experience early on in the disease.

Hypotesis and amis

Combining blood-based biomarkers, neuro-imaging, neuro-psychology and psychosocial factors (including caregiver experience), it could be possible to fill four major gaps: (i) scarce presence of scalable, non-invasive tools for very-early detection, (ii) the lack of a frameworks that capture the interaction of biological, psychological and social dimensions during the pre-clinical phases of AD, (iii) a superficial knowledge of how caregivers perceive and deal with AD in its various stages and (iv) the restricted knowledge of mutual influences between the experiences of the caregiver and of the patient.

Primary objectives are (PO.1) Jointly analyze biological, psychological, and social factors at different stages of the AD continuum to construct multidimensional clinical profiles and integrated risk models.

(PO.2) Examine the influence of psychological and social variables on the quality of life of patients and caregivers at different stages of the disease.

(Po.3) Investigate the relationship between caregiver psychological well-being and patient cognitive functioning, exploring potentially bidirectional relationships.

Secondary objectives are (SO.1) Compare biomarkers and neuropsychological performance at different stages of the AD clinical continuum.

(SO.2) Evaluate the diagnostic effectiveness of blood and neuroimaging biomarkers in discriminating the severity of cognitive impairment.

(SO.3) Explore stress and coping strategies adopted by caregivers, in relation to the stage of the disease and the quality of the dyadic relationship.

(SO.4) Integrate quantitative and qualitative data to understand the emotional experience of the caregiver throughout the entire disease continuum.

Ethical considerations

The study will be conducted in accordance with the ethical principles outlined in the Declaration of Helsinki, Good Clinical Practice (Legislative Decree 200/2007), and current regulations on the protection of personal data. In particular, the personal and sensitive data collected will be processed in compliance with Regulation (EU) 2016/679 (GDPR), Legislative Decree 196/2003, and the amendments introduced by Legislative Decree 101/2018. In order to guarantee the confidentiality of the data collected, all data will be pseudonymized by assigning an identification code (initials of the patient's surname and first name, as well as a consecutive number) that allows it to be stored and managed only by authorized personnel.

Sample

Consecutive outpatients, together with their respective caregivers, will be recruited at the Center for Cognitive Disorders and Dementias (CDCD) of ICS Maugeri IRCCS in Montescano, within the Neurophysiopathology Unit and the Diagnostic-Therapeutic Care Pathway for Dementia (DTCP). Patients may be either undergoing their first neurological evaluation for cognitive complaints or already followed by the Center for further diagnostic investigations aimed at the assessment of cognitive decline. Admission to the study will follow specific inclusion and exclusion criteria, which will be verified during the clinical evaluation. After determining the suitability of patients, the neurologist will offer them the opportunity to participate in the research, subject to signing the informed consent form and consent to the processing of personal data. Other imformation are reported in the eligibility section.

Procedure

All patients will undergo an initial clinical and neurological evaluation. Subsequently, routine blood tests will be performed to exclude secondary causes of cognitive impairment, along with structural neuroimaging investigations (magnetic resonance imaging or computed tomography) to rule out additional secondary causes and to assess cortical atrophy and cerebrovascular pathology. When clinically indicated, amyloid positron emission tomography (PET) will also be performed. Patients will then complete a standardized neuropsychological test battery assessing the main cognitive domains.

Based on the integration of these data, the neurologist will assign each patient to one of the following four diagnostic groups along the Alzheimer's disease continuum:

* Subjective Cognitive Decline (SCD): patients reporting subjective cognitive complaints in the presence of neuropsychological performance within normal limits.
* Mixed-etiology Mild Cognitive Impairment (MCI): patients with mild cognitive impairment not specifically attributable to Alzheimer's disease-related pathology.
* Alzheimer's disease-related Mild Cognitive Impairment: patients with mild cognitive impairment and a clinical-instrumental profile consistent with Alzheimer's disease pathology
* Early Alzheimer's disease: patients with mild dementia attributable to Alzheimer's disease.

After assignment to the clinical stage, when clinically appropriated, patients will undergo the assessment of plasma biomarkers of neurodegeneration and neuroinflammation. In addition, patients will complete a series of self-report questionnaires assessing emotional symptoms, perceived stress, quality of life, and cognitive reserve.

Concurrently with the patients' neuropsychological assessment, caregivers will be asked to complete selected self-report questionnaires evaluating caregiver burden, emotional symptoms, coping strategies, metacognitive beliefs, and quality of life. Furthermore, a subgroup of caregivers, selected through convenience sampling to ensure representation across the different patient clinical stages, will participate in a semi-structured interview conducted later.

ELIGIBILITY:
Inclusion Criteria (patients):

* Age ≥ 50 years.
* Presence of a primary caregiver, i.e., a person who provides regular care and who can actively participate in the study.
* Understanding of the research objectives and ability to provide informed consent.

Inclusion Criteria (caregivers):

* Be the primary caregiver, providing care for at least six months.
* Age ≥ 18 years, to ensure the ability to understand and actively participate in the study.
* Understanding of the research objectives and ability to provide informed consent.

Exclusion Criteria (patients):

* Age under 50.
* History of previous or concomitant neurological disorders (e.g., severe cerebrovascular accidents, brain tumors, traumatic injuries affecting cognitive functions) and neurodegenerative disorders.
* History of major psychiatric disorders (e.g., schizophrenia, severe bipolar disorder, untreated major depression), alcohol or substance abuse.
* Medical conditions that may interfere with cognitive function (e.g., advanced renal or hepatic failure, severe respiratory disorders, untreated hypothyroidism, B12 deficiency).
* Decompensated systemic diseases with clinical instability and significant organ failure.
* Marked sensory limitations (hearing or vision) and/or language difficulties.
* Participation in other experimental studies involving previous or current involvement in clinical trials of anti-amyloid drugs or experimental drug treatments for AD in the previous 6 months.

Exclusion Criteria (caregivers):

* Presence of severe active psychiatric disorders (e.g., untreated major depression, psychotic disorder, or schizophrenia).
* Difficulty participating in interviews and assessments due to language barriers, cognitive deficits, or other personal limitations.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatients and their caregivers will be enrolled at the Center for Cognitive Disorders and Dementia (CDCD) of the ICS Maugeri IRCCS in Montescano, within the Neurophysiopathology Unit and the diagnostic-therapeutic pathway for dementia (DTCP - Diagnostic-Therapeutic Care Pathway for Dementia).
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Mini Mental State Examination (MMSE) | Baseline
  This test is used for rapid screening of overall cognitive functioning. It consists of eleven items in different cognitive areas to obtain an overall score of cognitive functioning. Total scores range from 0 to 30 points. Lower scores indicate worse performances.
  N.B. This information will be collected only for the patients.
Montreal Cognitive Assessment (MoCA) | Baseline
  It is a cognitive screening test used in the assessment of dementia. The MoCA consists of several items that assess the following cognitive functions: visuospatial and executive functions, naming, attention, language, abstraction, memory, and spatial-temporal orientation. The score ranges from 0 to 30. Lower scores indicate worse performances.
  N.B. This information will be collected only for the patients.
Mental Deterioration Battery (MDB) | Baseline
  It is a battery of neuropsychological tests developed to assess cognitive decline, often used to diagnose and monitor cognitive disorders such as AD. The battery includes verbal memory tests (Rey's 15 words, immediate and delayed recall), phonemic verbal fluency, sentence construction, Raven's Progressive Matrices, immediate visual memory, freehand drawing copying, and programmed drawing copying. Each test is corrected independently. Lower scores indicate worse performances.
  N.B. This information will be collected only for the patients.
Free and Cue Selective Reminding Test (FCSRT) | Baseline
  is used to assess episodic memory and recall ability. The test consists of four main phases: learning phase, free recall, guided recall, and delayed recall. The final score is calculated by adding the scores from the different phases. Poor free recall but good guided recall suggests a retrieval deficit, which is compatible with normal aging. On the other hand, a low score in both conditions indicates memory consolidation difficulties.
  N.B. This information will be collected only for the patients.
Frontal Assessment Battery (FAB) | Baseline
  It is a test consisting of 6 items that measure conceptualization of similarity, lexical fluency in phonemic mode, motor planning, conflicting instructional responses, the go-no go task, and grasping behavior. Each item is scored on a scale from 0 to 3, with a maximum raw score of 18 points. Lower scores indicate worse performances.
  N.B. This information will be collected only for the patients.
Digit Span forward-backward | Baseline
  It is used to assess short-term verbal memory and verbal working memory. The test consists of two different tasks. The first task (forward) assesses short-term verbal memory and requires the assessor to read a sequence of numbers that the patient must then repeat in the same order. The second test (backward) assesses verbal working memory and requires the patient to repeat the sequence of numbers in reverse order to that read by the evaluator. The sequences gradually increase in difficulty, starting from a minimum of three digits up to a maximum of nine for the forward test and eight for the backward test. Lower scores indicate worse performances.
  N.B. This information will be collected only for the patients.
Span di cubi forward-backward | Baseline
  Psychometric tool used to assess short-term visuospatial memory and visuospatial working memory. The first test (forward) assesses short-term visuospatial memory and requires the evaluator to touch a sequence of cubes arranged on a board and the patient to repeat the sequence by touching the cubes in the same order. The second test (backward) assesses visuospatial working memory and requires the examiner to tap a sequence of cubes, which the patient must then repeat in reverse order. The sequences of cubes to be tapped gradually increase in difficulty, starting from a minimum of three cubes up to a maximum of nine for the forward test and eight for the backward test. Lower scores indicate worse performances.
  N.B. This information will be collected only for the patients.
Phonemic fluency | baseline
  It assesses vocabulary access and verbal fluency based on phonemic cues. It consists of three tests in which the patient must generate as many words as possible beginning with a specific letter (F, A, and S) in 60 seconds for each letter. The total raw score is the sum of the number of correct words generated for each letter within the time limit. Lower scores indicate worse performances.
  N.B. This information will be collected only for the patients.
Semantic fluency | Baseline
  Twop different test are included. Both assesse vocabulary access and verbal fluency on semantic prompts. Both consist of rials in which the patient must generate as many words as possible belonging to each of the following categories. For the first test categories are colors, animals, and fruits. instead, for the secon test categories are birds and pices of fornuture. The time allowed for each category is 60 seconds. The total raw score is the sum of the number of correct words generated for each letter within the time limit. Lower scores indicate worse performances.
  N.B. This information will be collected only for the patients.
Trail Making Test (TMT) A-B | Baseline
  A tool used to assess divided attention, visuomotor coordination, and the ability to alternate conceptual settings. Specifically, this test consists of two trials. Trial A (TMT-A) requires the patient to connect a list of randomly arranged numbers in ascending order as quickly as possible. Test B (TMT-B), on the other hand, requires the subject to connect alternating numbers and letters in the shortest possible time. The letters must be connected in alphabetical order and the numbers in ascending order. Shorter completion times indicate better performances.
  N.B. This information will be collected only for the patients.
Stroop test | Baseline
  It assesses selective attention and executive functions, with particular focus on inhibitory interference and cognitive flexibility. The test is divided into three parts of increasing difficulty. The first test consists of reading a list of colors. The second test requires the patient to name the color of the ink with which the circles are printed. Finally, in the third test, the patient is asked to name the color of the ink with which the names of the different colors are written. The patient is asked to try as quickly as possible and to continue the exercise even if they make mistakes. At the end, two raw scores are obtained: one for the completion time (with shorter completion times show better performances) and one for the number of mistakes made (with lower errors indicating a better performance)
  N.B. This information will be collected only for the patients.
Rey-Osterrieth Complex figure (ROCF) | Baseline
  This test consists of two different tasks. The first, ROCF copy, assesses visuospatial and motor planning skills. It consists of copying a complex figure as accurately as possible. The second test, or ROCF with 15-minute recall, assesses long-term visuospatial memory. Fifteen minutes after being shown a complex figure-a period during which the subject performs other non-interfering tasks-the subject is asked to reproduce the figure without being able to review it. For both of the trials, the total score is from o to 36. Lower scores indicate worse performances.
  N.B. This information will be collected only for the patients.
Multiple Features Target Target Cancellation | Baseline
  This test evaluates executive functioning. The patient is given a sheet containing a grid of visual stimuli, including both targets and distractors. They are then asked to cross out all the targets that correspond to the target stimulus. The execution time, the number of correctly identified targets, and the number of errors (number of distractors crossed out) are then recorded. These last two data points are then combined to calculate the accuracy index.
  Lower scores indicate worse performances.
  N.B. This information will be collected only for the patients.
Clock Drawing Test (CDT) | Baseline
  It is a brief neuropsychological screening tool used to assess global cognitive functioning, with particular sensitivity to executive functions, visuospatial abilities, attention, and planning. It includes three trials: a free-drawing condition, a pre-drawn circle condition, and a copy condition. Lower scores indicate worse performances.
  N.B. This information will be collected only for the patients.
Naming of colored photographs | Baseline
  It is a neuropsychological test used to assess lexical and semantic abilities, specifically object naming based on visual stimuli. The test consists of presenting a series of images depicting common objects, which the participant is required to name verbally. Lower scores indicate worse performances.
  N.B. This information will be collected only for the patients.
Episodic Memory Score | Baseline
  It is a composite index derived from standardized episodic memory tasks. It is designed to provide a synthetic and robust estimate of episodic memory functioning, reducing task-specific variability and enhancing sensitivity to early memory impairment. Lower scores indicate worse performances.
  N.B. This information will be collected only for the patients.
Semantic-Phonological Delta | Baseline
  It is a difference score calculated from verbal fluency tasks by subtracting phonological fluency performance from semantic fluency performance.
  This index captures the relative imbalance between semantic memory and executive-phonological processes. A reduced or negative delta reflects a disproportionate impairment in semantic fluency relative to phonological fluency.
  N.B. This information will be collected only for the patients.
Patient Health Questionnaire 9 (PHQ-9) | Baseline
  It is a psychological screening tool used to assess the severity of symptoms typical of major depressive disorder. The patient responds to the items by thinking about the frequency with which they have experienced the difficulties described in the last two weeks. Each item is rated on a 4-point Likert scale ranging from 0 (never) to 3 (almost every day). The total score, out of a maximum of 27 points, is given by the sum of the scores obtained for each item. Five levels of clinical severity have been identified, based on specific cut-offs: no depression (0-4 points), mild depression (5-9 points), moderate depression (10-14 points), moderately severe depression (15-19 points), and severe depression (20 or more points).
  N.B. This information will be collected both for patients and caregivers.
Generalized Anxiety Disorder (GAD-7) | Baseline
  It is a psychological screening tool used to assess the severity of symptoms typical of generalized anxiety disorder. It is a self-report questionnaire consisting of 7 items. The patient responds to the items by thinking about the frequency with which they have experienced the difficulties described in the last two weeks. Each item is rated on a 4-point Likert scale ranging from 0 (never) to 3 (almost every day). The total score, out of a maximum of 21 points, is given by the sum of the scores obtained for each item. Four levels of clinical severity have been identified, based on specific cut-offs: no anxiety (0-4 points), mild anxiety (5-9 points), moderate anxiety (10-14 points), and severe anxiety (15 or more points).
  N.B. This information will be collected both for patients and caregivers.
Perceived Stress Scale 10 (PSS-10) | Baseline
  It is a scale used to measure an individual's perceived stress level over the past four weeks. The aim is not to measure 20 specific areas, but rather the extent to which a person perceives their life as unpredictable or difficult to manage. The short version, in its Italian translation, has 10 items, each of which is rated on a 5-point Likert scale ranging from 0 (never) to 4 (very often). The total score (40 points) is given by the sum of the scores obtained for each item.
  N.B. This information will be collected both for patients and caregivers.
Metacognitions Questionnaire-30 (MCQ-30) | Baseline
  It is a self-report questionnaire consisting of 30 items, developed to assess metacognitive processes related to thought regulation and dysfunctional beliefs about mental functioning. It investigates five main metacognitive dimensions: (1) positive beliefs about worries; (2) negative beliefs about the uncontrollability and dangerousness of thoughts; (3) cognitive confidence; (4) need to control thoughts; (5) cognitive self-awareness. Each item is rated on a 4-point Likert scale from 1 (strongly disagree) to 4 (strongly agree), providing a total score and five subscores.
  N.B. This information will be collected both for patients (only those specifically selected according to their clinical diagnosis) and caregivers.
Cognitive Function Instrument self-report (CFI self-report) | Baseline
  This tool was created to assess patients' subjective perception of cognitive changes. It is useful for detecting and monitoring the early symptoms typical of neurocognitive disorders. The questionnaire consists of 14 items, each with three possible answers: yes (1 point), maybe (0.5 points), no (0 points). The final score (14 points) is given by the sum of the scores obtained for each item. The average reference score is 2.44±3.30. The higher the score obtained, the greater the cognitive difficulties self-perceived by the patient.
  N.B. This information will be collected only for the patients.
Cognitive Reserve Index Questionnaire short form (s-CRIq) | Baseline
  This is a tool designed to assess cognitive reserve. The questionnaire investigates three macro-aspects: education, occupation, and leisure activities. Four scores are obtained from the questionnaire: cognitive reserve index related to education level (CRI education), cognitive reserve index related to work experience (CRI work), cognitive reserve index based on leisure activities (CRI leisure), and overall cognitive reserve index calculated as the average of the three sub-indices (CRI). The scores are grouped into five different levels of cognitive reserve: low (points < 70), medium-low (71 < points < 84), medium (85 < points < 114), medium-high (115 < points < 130), and high (points > 130).
  N.B. This information will be collected both for patients and caregivers.
EuroQoL 5D e EuroQoL VAS | Baseline
  The EuroQoL 5d is a questionnaire that explores five different sections (mobility; personal care; usual activities; pain, discomfort, or distress; anxiety and depression) through various items that can be answered using a three-level Likert scale ranging from 1 (no problem) to 3 (severe problem). At the end of the administration, a 5-digit number is produced that represents the current and perceived quality of life. The EuroQoL VAS, on the other hand, is a visual analog scale that represents a graduated thermometer, whose temperature corresponds to the perceived quality of life. The scale ranges from 0 (worst possible health condition) to 100 (best possible health condition), and the respondent is asked to estimate their current level of health by marking the temperature that best represents it.
  N.B. This information will be collected both for patients and caregivers.
Multidimensional Assessment of Subjective Cognitive Decline (MASCoD) | Baseline
  It is a multidimensional screening tool designed to detect the memory and executive deficits that characterize SCD, helping to facilitate the differential diagnosis process and the identification of risk factors. The form includes a general section (aimed at collecting general clinical and sociodemographic information) and three specific sections. Section A (10 items) examines the main risk factors, comorbidities, and the possible presence of biomarkers. Section B (11 items) assesses subjectively perceived disturbances in memory and tasks involving attentional and executive functions. Finally, section C investigates the possible presence of psychological symptoms using items from the GAD-2 and PHQ-2. The total test score is given by the sum of the scores obtained in sections A and B (0-21). Three risk categories are identified: low risk (0-7 points), medium risk (8-13 points), and high risk (14-21 points).
  N.B. This information will be collected only for the patients.
Cognitive Function Instrument partner-report (CFI partner-report) | Baseline
  It is a tool created to assess a partner or caregiver's perception of a patient's cognitive difficulties. It is useful for identifying and monitoring early cognitive changes. The questionnaire consists of 14 items, each with three possible answers: yes (1 point), maybe (0.5 points), no (0 points). The final score (14 points) is given by the sum of the scores obtained for each item. The average reference score is 2.30±2.22. The higher the score obtained, the greater the cognitive difficulties found in the patient.
  N.B. This information will be collected only for the caregivers.
Caregiver Burden Inventory (CBI) | Baseline
  It is a questionnaire developed to measure the perceived burden of caregivers. It consists of 24 items organized into five subscales (objective time burden, developmental burden, physical burden, social burden, emotional burden). Each item is rated on a 5-point Likert scale with scores ranging from 0 (not at all) to 4 (extremely). The score (0-96) is higher the greater the perceived level of burden. Four levels of clinical severity have been identified, based on specific cut-offs: low burden (0-24), moderate burden (25-48), high burden (49-72), and very high burden (73-96). They are also analyzed separately to identify areas of greatest difficulty.
  N.B. This information will be collected only for the caregivers.
COPE NVI | Baseline
  It is a psychological questionnaire developed to assess the coping strategies used by a person to deal with stress. Specifically, it is a short Italian adaptation of the original version. It consists of 60 items that investigate coping strategies attributable to five main factors (avoidance, social support, positivity, problem solving, emotional distrust). Each item is rated on a 4-point Likert scale with scores ranging from 1 (I never do this) to 4 (I do this a lot). The score is calculated by adding up the responses for each subscale, providing a profile of the coping strategies adopted by the subject.
  N.B. This information will be collected only for the caregivers.
Instrumental Activity of Daily Living (IADL) | Baseline
  It is a scale used to assess the patient's level of independence in basic and instrumental activities of daily living. Eight complex functions are investigated (using the telephone, shopping, using transportation, cooking (only for women), doing housework (only for women), doing laundry (only for women), handling money, taking medication) and evaluated by assigning a score of 0 or 1. The total score is calculated by adding up the points assigned for each item. The maximum score varies between the two sexes. Specifically, it ranges from 0-8 for women and 0-5 for men. The higher the score, the greater the independence in basic daily instrumental activities.
  N.B. This information will be collected only for the caregivers.
Basic Activity of Daily Living (BADL) | Baseline
  It is a scale for assessing basic activities related to the patient's daily life. The scale investigates six activities (bathing; dressing; toileting; continence; moving around; eating) to which a score from 0 to 1 can be assigned (three alternatives in total, where two options share the same score, i.e., plausible alternatives that share the same level of severity). A score of 0 is assigned if the subject is dependent and a score of 1 if independent. The total score is calculated by adding up the points assigned for each item. The maximum score obtainable is 6, indicating total autonomy in activities of daily living.
  N.B. This information will be collected only for the caregivers.
Neuropsychiatric Inventory (NPI) | Baseline
  Developed to assess neuropsychological symptoms in patients with dementia or other neurological conditions. It investigates 12 neuropsychiatric domains (delusions, hallucinations, agitation/aggression, depression/dysphoria, anxiety, euphoria/excitement, apathy/indifference, disinhibition, irritability/lability, aberrant motor behaviors, sleep disturbances, eating disturbances), for each of which the presence or absence of the symptom must be noted. If the presence of the symptom is reported, its frequency (from 1=rarely to 4=very frequently) and severity (from 1=mild to 3=severe) must be assessed. Finally, the total score for the domain is calculated by multiplying the frequency by the severity. The total NPI score is obtained by adding the scores for all 12 domains (range 0-144). In general, scores between 0-10 indicate mild symptoms, between 11-30 moderate symptoms, and greater than 30 severe symptoms.
  N.B. This information will be collected only for the caregivers.
Family Strain Questionnaire-Short Form (FSQ-SF) | Baseline
  It is a screening tool designed to gather information on the situation experienced by a primary caregiver in the context of care. It consists of 30 items and a binary response scale (yes/no) and is particularly relevant for detecting psychological issues that warrant urgent, seriously recommended, recommended, or non-recommended psychiatric referrals/reports.
  N.B. This information will be collected only for the caregivers.
Semi-structured interview for caregivers | Baseline
  It will allow qualitative information to be gathered on the caregiver's experience in the daily management of patients with symptoms attributable to the AD continuum. It will aim to explore the burden of care, the perception of the disease, the emotional relationship between caregiver and patient, and the coping strategies adopted. In addition, future expectations and unmet needs will be explored. The interview questions will be organized according to a funnel approach, starting with more general aspects and then delving into more sensitive topics. Only a selected sub-sample of caregivers will participate in the interview.
  N.B. This information will be collected only for the caregivers.
Age of participants | Baseline
  Mean age of patients and caregivers assessed at study entry.
Sex distribution of participants | Baseline
  Number and percentage of patients and caregivers by sex.
Educational level of participants | Baseline
  Years of formal education completed by patients and caregivers.
Body Mass Index (BMI) | Baseline
  BMI calculated as weight in kilograms divided by height in meters squared (kg/m²).
Clinical and lifestyle characteristics | Baseline
  Number and percentage of participants presenting comorbidities, regular physical activity, tobacco use, alcohol consumption, and current medical therapy.
MRI or TC | Baseline
  In accordance with clinical guidelines, one of the following neuroimaging examinations will be performed to exclude secondary causes of cognitive impairment and to assess the presence of cortical atrophy and cerebrovascular disease.
  N.B. This information will be collected only for the patients.
Routine blood chemistry tests | Baseline
  In accordance with clinical guidelines, blood tests will be performed to exclude secondary causes of cognitive impairment.
  N.B. This information will be collected only for the patients.
Biomarkers of neurodegeneration and neuroinflammation | Baseline
  In a sample selected according to specific clinical criteria, plasma concentrations of blood biomarkers of neurodegeneration (Aβ40, Aβ42, p Tau181, and NfL) and blood biomarkers of neuroinflammation (GFAP, sTREM2, YKL40) will be analyzed.
  N.B. This information will be collected only for the patients.
Amyloid PET or FDG-PET | Baseline
  In a selected subgroup of patients, FDG-PET or amyloid PET will be performed based on diagnostic appropriateness and predefined clinical criteria. FDG-PET will be used to assess regional cerebral glucose metabolism as an index of neuronal dysfunction, while amyloid PET will be used to evaluate cerebral amyloid burden, supporting etiological characterization of cognitive impairment.
  N.B. This information will be collected only for the patients.

CONTACTS AND LOCATIONS:
Locations (1):
- ICS Maugeri Montescano Institute, Montescano, Pavia, Italy, Italy